CLINICAL TRIAL: NCT01916031
Title: Appropriate Care of URI (ACURI): Early Head Start
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Melissa Stockwell, MD, MPH, Asst Professor of Pediatrics and Population and Family Health, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: AAAD7081
Record Dates: First submitted 2013-08-01; First posted 2013-08-05 (Estimated); Last update posted 2013-08-05 (Estimated); Status verified 2013-08

CONDITIONS: Upper Respiratory Infection
MeSH Terms: conditions — Respiratory Tract Infections | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Education (Experimental): Upper Respiratory Infection education in Fall
  Interventions: Behavioral: Education
- Standard Curriculum (No Intervention)

INTERVENTIONS:
Behavioral: Education
  Arms: Education

SUMMARY:
The purpose of this study is to comparatively assess the effectiveness of a tailored educational intervention to improve health literacy levels regarding upper respiratory infections (URIs) and to decrease pediatric emergency department (PED) visits, among Latino households in Early Head Start.

ELIGIBILITY:
Inclusion Criteria:

* Attending an infant or toddler EHS group at participating site

Exclusion Criteria:

* Participant in pilot study
* Participant in community intervention regarding URI

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Number of pediatric emergency department visits | 5 months

SECONDARY OUTCOMES:
Use of over-the-counter medication | 5 months
Use of incorrect measuring tool | 5 months
Use of unprescribed antibiotic | 5 months
Knowledge regarding URI | 5 months
  Composite score

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Stockwell, MD MPH, Principal Investigator — Columbia University

REFERENCES:
- [Derived] Stockwell MS, Catallozzi M, Larson E, Rodriguez C, Subramony A, Andres Martinez R, Martinez E, Barrett A, Meyer D. Effect of a URI-related educational intervention in early head start on ED visits. Pediatrics. 2014 May;133(5):e1233-40. doi: 10.1542/peds.2013-2350. Epub 2014 Apr 7. PMID 24709931